CLINICAL TRIAL: NCT05538247
Title: Effects of Saccharomyces Boulardii CNCM I-745 on Intestinal Barrier Function
Brief Title: Saccharomyces Boulardii CNCM I-745 on Intestinal Barrier Function
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Michael Camilleri, MD, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 22-003898
Record Dates: First submitted 2022-09-08; First posted 2022-09-13 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Healthy
MeSH Terms: interventions — Indomethacin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- S. boulardii CNCM I-745 Group (Experimental): Subjects will receive Indomethacin from day 2 to day 7 and S. boulardii CNCM I-745 from day 1 to day 14
  Interventions: Drug: Indomethacin; Dietary Supplement: S. boulardii CNCM I-745
- Placebo Group (Placebo Comparator): Subjects will receive Indomethacin from day 2 to day 7 and Placebo from day 1 to day 14
  Interventions: Drug: Indomethacin; Drug: Placebo

INTERVENTIONS:
Drug: Indomethacin — Immediate release oral capsules 50 mg, 3 times a day for 6 days
Dietary Supplement: S. boulardii CNCM I-745 — Two 250 mg capsules orally twice daily for 14 days
  Other Names: Nonpathogenic yeast
  Arms: S. boulardii CNCM I-745 Group
Drug: Placebo — Two 250 mg capsules that contains no active study ingredient orally twice daily for 14 days
  Arms: Placebo Group

SUMMARY:
This study is being done to assess the effects of S. boulardii CNCM I-745 compared to placebo on impaired intestinal permeability, which is the control of material passing from inside the gastrointestinal tract through the cells lining the gut wall into the rest of the body.

DETAILED DESCRIPTION:
This placebo-controlled parallel group clinical study in healthy adults from the general population aims to investigate whether oral supplementation with S. boulardii CNCM I-745 could strengthen the intestinal barrier function and counteract the acute NSAID-induced hyperpermeability. Indomethacin will be used short term to increase intestinal permeability. The primary objective of the study is to assess the effects of S. boulardii CNCM I-745 on this impaired intestinal permeability.

ELIGIBILITY:
Inclusion Criteria:

* Considered as healthy after a comprehensive clinical assessment (detailed medical history and complete physical examination).
* With a body mass index (BMI) comprised between 18 and 35 kg/m^2 and weight > 50 kg at Screening.
* Able to comply with study requirements and to provide signed informed consent.
* Has signed the informed consent form before beginning any study procedure.
* Regular defecation (frequency and stool consistency, with at least about three bowel movements a week).
* For women of childbearing potential:

  * A negative urine pregnancy test immediately prior to starting the study treatment;
  * Agreement to comply with approved methods of contraception during the whole study: unless they meet the criteria of post-menopausal; i.e., 12 months of spontaneous amenorrhea, women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, including women whose career, lifestyle, or sexual orientation precludes intercourse with a male partner, should use one or more of the following acceptable methods of contraception that should be maintained throughout the study:
  * Surgical sterilization;
  * Hormonal contraception (implantable, patch, oral, intra-muscular);
  * Intra-uterine device;
  * Double barrier method (diaphragm plus condom);
  * At the discretion of the investigator, total abstinence is acceptable in cases where age, career, lifestyle, or sexual orientation of the patient ensures compliance.

Exclusion Criteria:

* History of hypersensitivity to the study treatments (active substance or excipients), brewer's or baker's yeast.
* Contraindication and special warning to the study treatments according to the Summary of Product Characteristics (SmPCs).
* History of chronic constipation with passage of fewer than 3 spontaneous bowel movements per week on average.
* History of chronic or recurrent diarrhea with spontaneous unformed bowel movements equivalent to or more often than 3 times daily.
* Prior gastrointestinal surgery (apart from appendectomy or cholecystectomy performed at least more than one year ago).
* History of Clostridium difficile infection.
* Active gastrointestinal disease.
* Known chronic or recurrent systemic disorder (including diabetes and hypertension) that may interfere with the study treatment evaluation.
* Associated immune deficiency.
* Severe hepatic or renal impairment.
* Clinically relevant abnormalities in results of laboratory tests as per Investigator's judgement.
* Patients with a central venous catheter.
* Oral or systemic antibacterial therapy during the 3 months prior to study enrollment.
* NSAIDs and proton pump inhibitor treatment longer than 1 week, within 3 months prior to study enrollment.
* Steroids within 6 weeks prior to study enrollment.
* Use of medications affecting gastrointestinal transit or permeability within 7 days prior to the testing.
* Use of artificial sweeteners, lactulose, mannitol within 2 days prior to the testing and during the 24 h testing period.
* New prescription medications during the 2 weeks prior to study enrollment.
* Use of probiotics or drugs that alters gut microbiota or function, during 4 weeks prior to study enrollment.
* Intake of antifungals within 14 days prior to study enrollment.
* Substantial changes in eating habits within 30 days prior to receiving the first dose of IMP product, as assessed by the Investigator.
* Current smoker.
* History or presence of drug or alcohol abuse.
* Inability to abstain from intensive muscular effort the day before the intestinal permeability test.
* Breast-feeding woman.
* Patients enrolled in another clinical trial within the past 30 days.
* Patients not able to fill in the study questionnaires.
* Any condition or personal circumstance that, in the opinion of the investigator, renders the subject unlikely or unable to comply with the full study protocol.

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2023-04-13 (Actual); Primary Completion 2025-12-30 (Actual); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Permeability assays | Baseline, 2 hrs, 8 hrs, 24 hours
  Change in intestinal permeability parameters urinary lactulose and 13C (13carbon) mannitol in 0-2 hrs, 2-8 hrs, 8-24 hr urine collection
Change in serum zonulin | Baseline, after intervention approximately 14 days
  Circulating zonulin will be measured by ELISA (Immundiagnostik AG) reported in ng/mL
Change in serum claudin | Baseline, after intervention approximately 14 days
  Serum Claudin 1, 2, 3, 4, 5 and 8 will be measured by ELISAs (Enzyme-Linked Immunosorbent Assay)
Change in fecal calprotectin | Baseline, day 7 (+/-1), day 14 (+/-1) and day 20 (placebo group only)
  Measured by ELISAs (Enzyme-Linked Immunosorbent Assay) from fecal samples reported in micrograms per milligram (μg/g)
Change in serum C-reactive protein (CRP) | Baseline, day 7 (+/-1), day 14 (+/-1) and day 20 (placebo group only)
  Measured by immuno-turbidimetric assay on an automated clinical chemistry analyzer reported in mg/L
Change in Gastrointestinal Symptom Rating Scale (GSRS) scores | Baseline, day 7 (+/-1), day 14 (+/-1) and day 20 (placebo group only)
  Measured by validated disease-specific questionnaire Gastrointestinal Symptom Response Scale (GSRS) used to evaluate common symptoms of gastrointestinal disorders. 15-item self-reported questionnaire related to signs and symptoms experienced by the subject during the past week, each rated on a seven-point Likert scale from no discomfort (score = 1) to very severe discomfort (score = 7). Total score is comprised between 15 and 105;

CONTACTS AND LOCATIONS:
Overall Officials: Michael Camilleri, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials